CLINICAL TRIAL: NCT04469491
Title: Treatment of COVID-19 by Nebulization of Inteferon Beta 1b Efficiency and Safety Study
Acronym: COV-NI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: CH TOURCOING (Unknown); CH ARROND DE MONTREUIL (Unknown); CH SAINT-QUENTIN (Unknown); CH Compiègne (Unknown); CH Abbeville (Unknown); CH VALENCIENNES (Unknown); Clinique Teissier (Unknown); University Hospital, Toulouse (Other); University Hospital, Angers (Other Government); CHU CAEN (Unknown); Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI2020_843_0041
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; INTERFERON; NEBULIZATION
Keywords: COVID-19; INTERFERON; NEBULIZATION
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled IFN arm (Experimental): IFN (Interferon) pulmonary (Inhalation) + routine care (+/- antibiotics; +/- dexamethasone; + appropriate O2 support)
  Interventions: Drug: inhaled type I interferon
- Control Arm: (Active Comparator): Aerosol (WFI water and routine care (+/- antibiotics;+/- dexamethasone; + appropriate O2 support).
  Interventions: Drug: WFI water nebulization

INTERVENTIONS:
Drug: inhaled type I interferon — The interventional arm includes inhaled interferon (9.6 MUI x2/d for 48 hours, then 9.6 MUI x1/d for 8 to 16 days or discharge), in addition to standard care. In phase B, maximum treatment duration is 8 days.
  Arms: Inhaled IFN arm
Drug: WFI water nebulization — The interventional arm includes a WFI water nebulization comparator.
  Arms: Control Arm:

SUMMARY:
COVID-19 is causing a serious viral pandemic in terms of health and social impact. To date, no treatment has yet demonstrated Strong efficacy in treating the infectious disease (COVID-19). Pulmonary administration of Interferon (IFN) type I is a therapeutic strategy with high potential,due to higher local concentrations and minimal adverse effects. Type I interferons (including IFN-α and IFN-β) are antiviral defence cytokines and also have the potential to negatively modulate IFN Type II and IL-6 dependent cytokine storm, the latter being induced in the late forms of COVID-19. In vitro, IFN-β were more effective on COVID-19 than IFN-α. In existing preliminary studies, only patients receiving IFN type I modulators have a decrease in viral carriage and a rapid reversal. The purpose of this project is to assess in hospitalized patients with oxygen for COVID 19, the clinical efficacy on oxygen requirements of the addition of inhaled Interferon type I compared to the control arm .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with laboratory-confirmed SARS-CoV-2 infection as determined by PCR < 96 h (at initial diagnosis or persistent carriage <96 h)
* Hospitalized patient with COVID-19 requiring oxygen therapy

And targeting in phase B :

* Patients under oxygen therapy such as nasal cannula/mask or non-invasive ventilation with paO2/FiO2 > 200 mmHg.
* Patients hospitalized for less than 7 days.
* Patients with symptoms for less than 10 days or RT-PCR (<96h) with Cycle Treshold < 25.
* Social security coverage
* signed informed consent (by patient or their legally authorized representative)

Exclusion Criteria:

* Hypersensitivity to natural or recombinant interferon-ß
* Hypersensitivity to human albumin or mannitol
* Recent suicide attempt
* Decompensation of liver failure
* age < 18 years
* Pregnant or nursing.
* Patients managed on an outpatient basis (i.e. not initially hospitalized).
* Parenteral IFN treatment. In periode B, addition of new exclusion criteria
* Patients with kidney transplant
* Immunocompromised patients
* Patients with severe systemic disease constantly threatening their vital prognosis (ASA ≥ IV: e.g. severe ARF, advanced cancer pathology, recent myocardial IDM, severe valvular dysfunction, dependence on parenteral nutrition on central line, shock, sepsis, trauma, ...).
* Patients in septic shock.
* Patients with documented fungal infection.
* Patients on mechanical ventilation.
* Patients hospitalized for COVID-19 for more than 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
oxygen requirement score at day 0 | day 0
  oxygen requirement score at day 0
oxygen requirement score at day 15 | day 15
  oxygen requirement score at day 15
Variation oxygen requirement score between day 0 and day15 | at day 15
  Variation oxygen requirement score between day 0 and day15

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lanoix, MD, Principal Investigator — CHU Amiens
Locations (7):
- France (7):
  - CH d'Abbeville, Abbeville
  - CHU Amiens, Amiens
  - CH Compiègne-Noyon, Compiègne
  - CH de l'Arrondissement de Montreuil-sur-mer, Rang-du-Fliers
  - CH de Saint-Quentin, Saint-Quentin
  - CH de Tourcoing, Tourcoing
  - CH de valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No